CLINICAL TRIAL: NCT02030431
Title: Dynaloc vs. Multiple Cancellous Screws for Treatment of Femoral Neck Fractures
Brief Title: Dynaloc for Treatment of Femoral Neck Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: overweight of hard-ware removals in the Dynaloc group
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Lars C. Borris, Consultant of Orthopaedic surgery, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-362-13
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cancellous screws (Active Comparator): Patients in this group are having osteosynthesis with three screws
  Interventions: Device: Cancellous screws
- Dynaloc (Active Comparator): Patients in this group are having osteosynthesis with Dynaloc (three screws fixed in a small plate)
  Interventions: Device: Dynaloc

INTERVENTIONS:
Device: Dynaloc
  Arms: Dynaloc
Device: Cancellous screws
  Arms: Cancellous screws

SUMMARY:
A prospective, randomized study comparing the effectiveness of a new system, Dynaloc compared with three cancellous screws, for osteosynthesis of femoral neck fractures

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (see age specifications below) with subcapital femoral neck fractures (stable or unstable) confirmed with anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Patients between 50 and 69 years of age with any Garden type femoral neck fracture
* Patients older than 70 years of age with femoral neck fractures Garden type I and II
* Patients older than 70 years of age with a femoral neck fracture Garden types III and IV and contraindication to hemiarthroplasty.
* Operative treatment within 4 days (i.e., 72 hours) of presenting to the emergency room.
* Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
* Anticipated medical optimalization of the patient for operative fixation of the hip.
* Provision of informed consent by patient or proxy.
* Low energy fracture (defined as a fall from standing height).
* No other major trauma.

Exclusion Criteria:

* Associated major injuries of the lower extremity (i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture).
* Retained hardware around the affected hip.
* Abnormal opposite hip making end-point evaluation impossible
* Infection around the hip (i.e., soft tissue or bone).
* Patients with disorders of bone metabolism other than osteoporosis (i.e., Paget's disease, renal osteodystrophy).
* Moderate or severe cognitively impaired patients (i.e., Six Item Screener with three or more errors).
* Patients with Parkinson's disease (or dementia or other neurological deficit) severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation.
* Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Shortening of the femoral neck | 1 year

SECONDARY OUTCOMES:
Reoperation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark